CLINICAL TRIAL: NCT04013945
Title: A Randomised, Double-blinded, Parallel, Placebo-controlled Study to Investigate the Effect of Superba Boost (Krill Oil Concentrate) on Various Skin Parameters in Healthy Adult Subjects.
Brief Title: Study to Investigate the Effect of Superba Boost on the Skin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aker BioMarine Human Ingredients AS (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AFCRO-097
Record Dates: First submitted 2019-07-06; First posted 2019-07-10 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Physiology, Skin
MeSH Terms: interventions — Exercise; Plant Oils

STUDY DESIGN:
Intervention Model Description: Subjects who successfully meet the eligibility criteria will be randomized on a 1:1 basis, to receive Superba Boost or Placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be carried out by computer-generated block-randomization lists. Subjects will be randomized to one of the two treatment groups, in blocks of 6. The randomization will be seeded, with the seed only available to the statistician generating the randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Superba Boost capsules (Active Comparator): 1000 mg krill oil concentrate per capsule
  Interventions: Dietary Supplement: Superba Boost (Active)
- Placebo capsules (Placebo Comparator): 1000 mg capsule composed of mixed vegetable oil.
  Interventions: Dietary Supplement: Vegetable oil (Placebo)

INTERVENTIONS:
Dietary Supplement: Superba Boost (Active) — To assess changes in Trans-epidermal water loss (TEWL), measured at baseline and after 12 weeks of daily consumption with Superba Boost.
  Arms: Superba Boost capsules
Dietary Supplement: Vegetable oil (Placebo) — To assess changes in Trans-epidermal water loss (TEWL), measured at baseline and after 12 weeks of daily consumption with Placebo.
  Arms: Placebo capsules

SUMMARY:
Study to determine the effect of 12 weeks daily consumption of Superba Boost as compared to placebo on changes in Trans-Epidermal Water-Loss (TEWL).

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel group trial in 70 healthy adult male and female subjects between 20 and 50 years. The primary objective is to assess whether Superba Boost krill oil administered at a dose of 1 g per day for 12 weeks (84 days) has a positive effect on the TEWL, skin hydration and elasticity. At screening, the subjects must have TEWL values of >10 g/m2/h and <24.9 g/m2/h when measured by a TEWAmeter, i.e. within the range defined as normal and healthy skin. The change in omega-3 index, defined as EPA and DHA as percentage of total fatty acids in red blood cells, will be measured and correlated to the changes in the skin parameters.

The study consists of 4 visits: the screening visit (V1), baseline visit / week 0 / Start of treatment (V2), Interim / Week 6 (V3) and week 12 / end of treatment (V4) . In this study, subjects must have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less will be recruited. Each subject must fulfill all inclusion criteria and will not be allowed to meet any of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, the subject must fulfil all of the following criteria:

* Be able to give written informed consent;
* Be aged between 20 and 50 years, inclusive;
* Trans-epidermal water loss score >10 and ≤ 24.9 g/m²/h;
* Be in general good health with no existing co-morbidities
* Have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less;
* Be willing to avoid all fish and seafood meals in the 4-days before each scheduled clinic visit;
* Be willing to maintain dietary habits and physical activity levels throughout the trial period;
* Be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the Investigator;
* Willing & able to consume the investigational product daily for the duration of the study.

Exclusion:

The presence of any of the following criteria will exclude the subject from participating in the study:

* Pregnant or breastfeeding women; women planning to become pregnant during the study;
* Women of child-bearing potential who do not use an acceptable method of contraception;
* Suffer from photosensitivity;
* History of skin cancer;
* Are currently taking photosensitizing medication, or have done so in the previous 4 weeks;
* Sunbed tanning or sunbathing in preceding 3 months, or planned sunbed tanning or sunbathing during the study period
* Taking supplements known to have an effect on skin (e.g. fish oil, coenzyme Q-10, garlic, lycopene, beta-carotene, etc.), or have done so in the previous 4 weeks, except for medically-prescribed supplements or natural health products.
* Supplements known not to have an effect on the skin (e.g. probiotics) are allowed, once the subject has been on a stable dose for greater than 3 months and are willing to continue this supplement for the duration of the study;
* Systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg. Subjects receiving blood pressure medications, must be on stable dose for greater than 3 months;
* Known allergy to seafood;
* Are hypersensitive to any of the components of the test product;
* Disturbed absorption due to changes in the gastrointestinal tract (e.g., resections, diverticula, malabsorption, blind-loop syndrome);
* Known alcohol abuse (> 21 units of alcohol per week) or drug abuse within the previous year of screening;
* Clinically significant illness within 14 days prior to dosing;
* Current or recent (within 3 months of screening visit) changes in diet, which in the opinion of the Investigator, deviates from a normal diet (e.g. vegetarians may be acceptable, vegans are not acceptable);
* Planned major changes in life style (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
* Has any health conditions that would prevent from fulfilling the study requirements, put the subject at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results;
* Are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year);
* Experiences alarm features such as weight loss, rectal bleeding, recent change in bowel habit (<3 months) or abdominal pain;
* Have a malignant disease or any concomitant end-stage organ disease;
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
* Subjects receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
12 weeks daily consumption of Superba Boost as compared to placebo on changes in Trans-Epidermal Water-Loss (TEWL) will be measured. | 12 weeks.
  Trans-epidermal water loss (the loss of water that passes from inside the body through the skin to outside the body) measured at baseline and after 12 weeks of intervention using a TEWAMetre will be considered. This measurement provides information on the integrity of the skin protective barrier functions. Subjects eligible for the study will have a TEWL value >10 and ≤ 24.9 g/m²/h. In comparison, A TEWL value between 0-9 is classified as a "very healthy" barrier function and values between 25-34 are in the "strained" range. These participants will therefore be deemed ineligible for the study. Additionally, subjects with a TEWL value of >35 will have a skin barrier function classified as "critical" and will also be ineligible for the study.

SECONDARY OUTCOMES:
Daily consumption of Superba Boost as compared to placebo on changes of in TEWL values. | 12 weeks.
  The effect of daily consumption of Superba Boost as compared to placebo on changes in Trans-Epidermal Water-Loss (TEWL) from baseline to 6 weeks after start of treatment, and from 6 weeks of treatment to the end-of-study will be measured.
The effect of daily consumption of Superba Boost as compared to placebo on changes in skin hydration will be measured. | 12 weeks.
  The effect of daily consumption of Superba Boost as compared to placebo on changes in skin hydration from baseline (pre-study) to 6 weeks after start of treatment, and from 6 weeks of treatment until end-of-study will be considered. The Corneometer indicates the hydration level of the top layers of the skin. The value of the dielectric constant is directly proportional to the level of skin hydration. i.e. higher value= more hydrated skin. The measurements for skin hydration are as follows: 0-29.9 (Very Dry), 30-44.9 (Dry), 44-130 (Normal).
The effect of daily consumption of Superba Boost as compared to placebo on changes in skin firmness will be measured. | 12 weeks.
  The effect of daily consumption of Superba Boost as compared to placebo on changes in skin firmness from baseline (pre-study) to 6 weeks after start of treatment, and from 6 weeks of treatment until end-of-study will be considered. The Cutometer measures the resistance of the skin to be sucked up by negative pressure (firmness) and its ability to return into its original position (elasticity). Elasticity is measured from 0 (no elasticity) to 1 (maximum elasticity).
The effect of daily consumption of Superba Boost as compared to placebo on subjective evaluation by study subjects, using questionnaires will be studied. | 12 weeks.
  The effect of daily consumption of Superba Boost as compared to placebo on subjective evaluation by study subjects, using questionnaires, after 6 and 12 weeks of treatment will be considered. Subjects will be provided with a "Subject Skin Evaluation" Questionnaire and will answer questions regarding "Overall Skin Condition", "Skin Hydration", "Skin Moisture" and "Skin Elasticity and Firmness" of their own skin. Changes in the subjects' interpretation of their own skin condition will therefore be reported over the 12-week study period.
  Each subject reports their opinion of their own skin condition through a numeric scale measuring from 0 to 100mm. 0mm is the "worst" skin condition and 100mm is the "best".
The effect of daily consumption of Superba Boost as compared to placebo on Omega-3 index will be measured. | 12 weeks.
  The effect of daily consumption of Superba Boost as compared to placebo on Omega-3 index, using a blood spot collected by fingerpick will be considered. The higher the percentage (%), the higher the Omega-3 content of the blood.

OTHER OUTCOMES:
Depending on the outcome of the primary and secondary objectives, further exploratory analysis may be performed on the skin samples to meaure the effect of Superba Boost versus the placebo on the Lipid content of skin | 12 weeks.
  Analysis will be performed on the following lipids: Nonhydroxydehydrosphingosine (NdS), Nonhydroxysphingosine (NS), Nonhydroxyphytosphingosine (NP), Nonhydroxy-6-hydroxysphingosine (NH), Alphahydroxydehydrosphingosine (AdS), Alphahydroxysphingosine (AS), Alphahydroxyphytosphingosine (AP), Alphahydroxy-6-hydroxysphingosine (AH), Omegahydroxysphingosine (EOS), Omegahydroxyphytosphingosine (EOP), Omegahydroxy-6-hydroxysphingosine (EOH), Omegahydroxydehydrosphingosine (EOdS)); diacylglycerol; free cholesterol; cholesterol esters; triacylglycerols. In the case of all the above lipids, the higher the percentage (%), the higher the lipid content of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Aoife Hayes, PhD, Study Director — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food CRO, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No